CLINICAL TRIAL: NCT05602831
Title: Using Peripheral Blood Circulating Tumor DNA (ctDNA) Based Human Papillomavirus (HPV) and Genetic Variant Test to Assess the Prognosis of Surgery or Radical Chemoradiotherapy in Patients With Locally Advanced Cervical Cancer
Brief Title: Assessment of Prognosis Using Peripheral Blood Circulating Tumor DNA in Patients With Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Amoy Diagnostics (Industry)
Responsible Party: Principal Investigator, Xiaohua Wu MD, Director of Gynecologic Oncology, Fudan University
Other Study IDs: LACC-BD-1
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Locally Advanced Cervical Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue and peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- operable treatment group: After enrollment, patients will receive standard treatment and conventional follow-up strategy.
  Peripheral blood samples will be collected before treatment and at different time points after starting treatment.
  Baseline surgical tissue will be also obtained.
  Interventions: Other: detect HPV and genetic variants
- radical chemoradiotherapy group: After enrollment, patients will receive standard treatment and conventional follow-up strategy.
  Peripheral blood samples will be collected before treatment and at different time points after starting treatment.
  Baseline puncture tissue will be also obtained before radical chemoradiotherapy.
  Interventions: Other: detect HPV and genetic variants

INTERVENTIONS:
Other: detect HPV and genetic variants — Serum tumor markers and ctDNA HPV and genetic variants will be detected in peripheral blood samples. HPV and genetic variants will be also detected in baseline surgical tissues.
  Groups: operable treatment group
Other: detect HPV and genetic variants — Serum tumor markers and ctDNA HPV and genetic variants will be detected in peripheral blood samples. HPV and genetic variants will be also detected in baseline puncture tissues.
  Groups: radical chemoradiotherapy group

SUMMARY:
This observational study is conducted to assess the value of using peripheral blood ctDNA to detect dynamic changes in HPV and genetic variants in predicting the prognosis of patients with locally advanced cervical cancer, as compared with traditional imaging and tumor markers.

DETAILED DESCRIPTION:
The goal of this study is to assess the prognostic value of ctDNA HPV and gene variant clearance in peripheral blood.

Two cohorts will be enrolled: operable group and radical chemoradiotherapy group.

After enrollment, patients will receive standard treatment and follow-up strategy. Peripheral blood samples will be collected from 2 cohorts of patients before treatment and at different time points after starting treatment. Baseline surgical or puncture tissues will be also obtained.

Peripheral blood ctDNA and baseline tissues will be tested for HPV copy number based on ddPCR and genetic variation based on next-generation sequencing (NGS).

Finally, the correlation of ctDNA HPV and genetic variation clearance with patients prognosis and its value for recurrence monitoring compared to traditional tumor markers and imaging examination will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial diagnosis, operable locally advanced cervical cancer, FIGO stage IB2/3-IIA1/2 or initial diagnosis, receive radical chemoradiotherapy locally advanced cervical cancer, FIGO stage IIB-IVA
* Not receiving systemic treatment
* Pathological diagnosis: cervical squamous cell carcinoma
* Aged 18-70 years
* ECOG PS: 0-1
* Patients volunteer to participate in this study and sign the informed consent, with good compliance, and cooperate with the acquisition of tissue samples and blood samples

Exclusion Criteria:

* Patients diagnosed with other malignancies within 5 years
* Patients had received previous systemic antitumor therapy
* In the judgment of the investigator, the patients had other factors that might have caused the study to be discontinued

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A：Patients with initial diagnosis, operable locally advanced cervical cancer, FIGO stage IB2/3-IIA1/2.
  Cohort B：Patients with initial diagnosis, receive radical chemoradiotherapy locally advanced cervical cancer, FIGO stage IIB-IVA.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Two years
  Assess PFS in ctDNA HPV and genetic variants clearance versus not clearance

SECONDARY OUTCOMES:
Overall Survival (OS) | Two years
  Assess OS in ctDNA HPV and genetic variants clearance versus not clearance
Recurrence prediction performance of ctDNA dynamic changes | Two years
  Performance of dynamic changes of HPV copy number and genetic variation in ctDNA in predicting recurrence compared with imaging and serum tumor markers

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No